CLINICAL TRIAL: NCT03599687
Title: Soiled Airway Tracheal Intubation and the Effectiveness of Decontamination by Paramedics (SATIATED): A Randomised Controlled Manikin Study
Brief Title: Soiled Airway Tracheal Intubation and the Effectiveness of Decontamination by Paramedics
Acronym: SATIATED
Status: Completed | Type: Observational
Sponsor: Yorkshire Ambulance Service NHS Trust (Other Government)
Collaborators: College of Paramedics (Unknown)
Responsible Party: Sponsor
Other Study IDs: YASRD100; 245954 (Other: IRAS)
Record Dates: First submitted 2018-07-12; First posted 2018-07-26 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Airway Management; Intubation, Intratracheal; Laryngoscopy; Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Training in SALAD technique — The training session will be delivered, and will take around 45 minutes to complete, including time for participant practice. The training intervention will adopt the Advanced Life Support Group/Resuscitation Council 4-stage approach of skills teaching, and is comprised of: A real-time demonstration of the SALAD technique by the researcher; A repeated demonstration with an explanation of the rationale of the steps taken when performing SALAD (not real-time); Another demonstration of the SALAD technique conducted by the researcher, but guided by one of the participants; An attempt by the same participant who guided the researcher in the previous step, followed by a practice attempt by the other participants.

SUMMARY:
In more than one-in-five cases of out-of-hospital cardiac arrest, airways are blocked by vomit and blood. Sometimes, paramedics cannot clear the airway using methods they have been taught. If the airway cannot be cleared, the patient will die.

Usually, these patients will have a breathing tube placed into their windpipe (intubation), as this provides protection from vomit and blood. To do this, the paramedic needs to be able to see the entrance to the windpipe.

A new method of clearing the airway called SALAD has been used in patients to help insert a breathing tube, but it is not known whether the method can help paramedics. This study will use a manikin to see if paramedics can insert a breathing tube more often on their first attempt, using SALAD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* HCPC registered paramedic employed by Yorkshire Ambulance Service
* Authorised to intubate within Yorkshire Ambulance Service
* No SALAD training in the last 3 months

Exclusion Criteria:

* Not an HCPC registered paramedic employed by Yorkshire Ambulance Service
* Not authorised to intubate within Yorkshire Ambulance Service
* Allergy to artificial 'vomit' ingredients
* Unwilling to provide consent
* SALAD training in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be NHS staff who are employed by Yorkshire Ambulance Service NHS Trust, and who are Health and Care Professions Council (HCPC) registered paramedics.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pilbery, Principal Investigator — Yorkshire Ambulance Service NHS Trust
Locations (1):
- Yorkshire Ambulance Service NHS Trust, Wakefield, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Group AAB: In order to adjust for improvements in participant performance that might arise from repeated attempts at intubation, beyond that of the SALAD training itself, paramedics were randomised into one of two group. In AAB, participants randomised into making two pre-training and one post-training intubation attempts.
- Group ABB: Participants randomised into making one pre-training and two post-training intubation attempts.
Period: Overall Study
Arm/Group | Group AAB | Group ABB
Started | 82 | 82
Completed | 82 | 82
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group AAB | Group ABB | Total
Number analyzed (Participants) | 82 | 82 | 164
Age, Customized [Count of Participants; unit: Participants]
  Adults > 18 years | 82 | 82 | 164
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Unknown | 82 | 82 | 164
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 82 | 82 | 164
Intubation attempts in past 12 months [Median (Inter-Quartile Range); unit: attempts] | 2.5 [0 to 6] | 3.0 [1 to 7] | 3.0 [1 to 6.5]
Successful intubation attempts in past 12 months [Median (Inter-Quartile Range); unit: attempts] | 2 [0 to 5] | 2 [0 to 6] | 2 [0 to 6]
Years as a paramedic [Median (Inter-Quartile Range); unit: years] | 5 [1 to 10] | 3.5 [0 to 10] | 4 [1 to 10]
Awareness of SALAD technique [Count of Participants; unit: Participants] | 15 | 21 | 36

OUTCOME MEASURES:

1. Primary Outcome: Difference in First-pass Intubation Success Rates Before and After SALAD Training
Description: This measure is a comparison of Group AAB's first-pass intubation success rate, using an attempt which occurred before SALAD training, and Group ABB's intubation success rate, using an intubation attempt that occurred after SALAD training.
Time Frame: pre- and post-training as part of 2 hour study session
Measure: Count of Participants; unit: Participants
Arm/Group | Group AAB | Group ABB
Number analyzed (Participants) | 82 | 82
Participants | 44 | 74

2. Secondary Outcome: Difference Between Mean Time Taken (in Seconds) to Perform a Successful Intubation on the First- Attempt, Before and After SALAD Training Approximately 30 Minutes Apart.
Time Frame: seconds
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Group AAB | Group ABB
Number analyzed (Participants) | 23 | 28
seconds | 15.4 (3.5) | 3.7 (3.4)

3. Secondary Outcome: Difference in Success Rates Between Participants Who Have Two Post-training Intubation Attempts Versus Participants Who Only Have One Post-training Intubation Attempt
Time Frame: pre- and post-training as part of 2 hour study session
Measure: Count of Participants; unit: Participants
Arm/Group | Group AAB | Group ABB
Number analyzed (Participants) | 82 | 82
Participants | 71 | 73

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the course of each study session, which lasted approximately 2 hours.
Description: Adverse events are reported to the service via the DATIX incident reporting scheme and the sponsor is notified immediately.
Arm/Group | Group AAB | Group ABB
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/82
Other Adverse Events (participants affected / at risk) | 0/82 | 0/82

LIMITATIONS AND CAVEATS:
Manikin study Vomit did not contain solid material and was not odorous Participants not blinded from allocation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT03599687/Prot_SAP_000.pdf